CLINICAL TRIAL: NCT07242209
Title: The Relationship Between Menstrual Cycle Phases and Postoperative Nausea and Vomiting: The Role of Sugammadex
Brief Title: Sugammadex and Menstrual Cycle in Postoperative Nausea and Vomiting
Status: Recruiting | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burçin Alaçam, MD, Anesthesiology Specialist, Sakarya University
Other Study IDs: E-43012747-050.04-513202-482
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Nausea and Vomiting; Menstrual Cycle
Keywords: postoperative nausea and vomiting; menstruel cycle; septorhinoplasty; sugammadex; female reproductive age
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group Follicular: Women in the follicular phase of their menstrual cycle undergoing septorhinoplasty.
  Interventions: Other: PONV Assessment Questionnaire
- Group ovulatory: Women in the ovulatory phase of their menstrual cycle undergoing septorhinoplasty.
  Interventions: Other: PONV Assessment Questionnaire
- Group Luteal: Women in the luteal phase of their menstrual cycle undergoing septorhinoplasty.
  Interventions: Other: PONV Assessment Questionnaire

INTERVENTIONS:
Other: PONV Assessment Questionnaire — All participants will complete a standardized postoperative questionnaire designed to assess the presence, frequency, and severity of nausea and vomiting within the first 24 hours after septorhinoplasty surgery. The questionnaire will be administered in the post-anesthesia care unit and during the postoperative follow-up period. Responses will be recorded by trained research staff or anesthesia team members. No experimental drug or additional therapeutic intervention will be applied. The collected data will be used to evaluate possible associations between postoperative nausea and vomiting (PONV) incidence and the menstrual cycle phase (follicular, ovulatory, or luteal). In addition, anesthetic records will be reviewed to document the use of routinely administered perioperative agents, including sugammadex, to assess their potential influence on PONV outcomes.

SUMMARY:
This observational study aims to evaluate the relationship between menstrual cycle phases and the incidence of postoperative nausea and vomiting (PONV) in women of reproductive age undergoing septorhinoplasty surgery. The study's primary objective is to determine whether different phases of the menstrual cycle are associated with variations in PONV frequency. As a secondary objective, the relationship between menstrual phases, PONV incidence, and the use of sugammadex during anesthesia will be analyzed. No additional intervention will be applied beyond routine clinical practice; all data will be collected prospectively from anesthesia records and postoperative evaluations.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effect of menstrual cycle phases on the incidence of postoperative nausea and vomiting (PONV) in women of reproductive age undergoing septorhinoplasty under general anesthesia. PONV is a common postoperative complication that can negatively impact patient recovery, prolong discharge time from the post-anesthesia care unit, and decrease overall patient satisfaction. Several risk factors for PONV have been identified, and recent consensus guidelines published in 2020 have also suggested that the menstrual cycle may influence PONV risk.

In this prospective observentional study, participants will be randomly assigned to receive either preoperative nebulized lidocaine or nebulized 3% sodium chloride solution, administered 15 minutes before surgery. The primary objective is to determine whether menstrual cycle phase (follicular, ovulatory, or luteal) is associated with differences in PONV incidence. The secondary objective is to evaluate whether the use of sugammadex during anesthesia has an additional effect on PONV occurrence across different menstrual phases.

Sugammadex, a modified γ-cyclodextrin that selectively binds aminosteroidal neuromuscular blocking agents such as rocuronium, may also interact with endogenous steroid hormones. Pharmacokinetic studies have shown that sugammadex exposure can decrease progesterone levels by approximately 34% and may reduce estrogen levels as well. Given the hormonal fluctuations during the menstrual cycle, understanding these interactions may help identify specific phases associated with increased PONV risk and support the development of individualized anesthesia management strategies.

All participants will receive standard anesthetic and surgical care. PONV assessment will be performed in the postoperative care unit and during the first 24 hours after surgery. Demographic data, anesthetic drug information, menstrual cycle phase, and PONV outcomes will be recorded and statistically analyzed.

The results of this trial may contribute to improved understanding of the interaction between hormonal status, anesthetic drugs, and postoperative outcomes, potentially informing future preventive measures for PONV in women undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age between 18 and 40 years
* Regular menstrual cycle
* Scheduled for ENT (ear, nose, and throat) surgery
* Classified as ASA physical status I or II

Exclusion Criteria:

* Irregular menstrual cycle
* Unknown date of last menstrual period
* Receiving estrogen and/or progesterone supplementation
* Pre-menopausal or menopausal status
* Pregnant
* Breastfeeding
* Classified as ASA physical status III or IV
* Apfel score ≥ 3
* History of drug allergy
* Surgery duration exceeding 3 hours
* Age <18 or >40 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: The study population consists of women of reproductive age (18-40 years) who are scheduled to undergo septorhinoplasty surgery under general anesthesia. Eligible participants have a regular menstrual cycle and are classified as ASA physical status I or II. Participants with irregular menstrual cycles, unknown last menstrual period, pre-menopausal or menopausal status, or those receiving hormonal supplementation are excluded. Other exclusion criteria include pregnancy, breastfeeding, ASA III-IV status, high risk for postoperative nausea and vomiting (Apfel score ≥3), history of drug allergy, and surgery duration exceeding 3 hours. Data will be collected prospectively from anesthesia records, postoperative assessments, and standardized questionnaires evaluating postoperative nausea and vomiting (PONV).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | Within 24 hours after surgery
  The primary outcome of this study is the incidence of postoperative nausea and vomiting (PONV) within the first 24 hours after septorhinoplasty surgery. PONV will be evaluated using a standardized questionnaire administered during the postoperative recovery period and at 24 hours post-surgery. The presence, frequency, and severity of nausea and vomiting will be recorded. Data will be analyzed according to the menstrual cycle phase (follicular, ovulatory, luteal) to determine possible associations between menstrual phase and PONV occurrence.

SECONDARY OUTCOMES:
Relationship Between Sugammadex Use and Postoperative Nausea and Vomiting (PONV) | 24 hours after surgery
  This outcome evaluates whether the use of sugammadex during anesthesia is associated with the incidence of postoperative nausea and vomiting (PONV) in women undergoing septorhinoplasty. Anesthetic records will be reviewed to determine sugammadex administration and dosage. PONV incidence within the first 24 hours postoperatively will be compared between patients who received sugammadex and those who did not.
Relationship Between Sugammadex Use and Menstrual Cycle Phase | During anesthesia administration in surgery
  This outcome evaluates whether sugammadex administration during anesthesia is associated with the menstrual cycle phase in women undergoing septorhinoplasty. Anesthetic records will be reviewed to determine sugammadex use, and menstrual cycle phase (follicular, ovulatory, luteal) will be recorded. The analysis aims to explore potential interactions between sugammadex exposure and hormonal variations across the menstrual cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University-Anesthesiology and Reanimation Department, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study will not share individual participant data. Data will be collected and analyzed solely for research purposes and will remain confidential in accordance with institutional and ethical guidelines.

REFERENCES:
- [Result] Sener EB, Kocamanoglu S, Cetinkaya MB, Ustun E, Bildik E, Tur A. Effects of menstrual cycle on postoperative analgesic requirements, agitation, incidence of nausea and vomiting after gynecological laparoscopy. Gynecol Obstet Invest. 2005;59(1):49-53. doi: 10.1159/000081222. Epub 2004 Sep 30. PMID 15467297